CLINICAL TRIAL: NCT04794166
Title: Do Lumbar Spine Surgery Patients With Dura Rupture Differ in Symptom Prevalence and Severity From Other Lumbar Spine Surgery Patients in the Early Postoperative Phase
Brief Title: Symptom Prevalence and Severity in Lumbar Spine Surgery With and Without Dura Rupture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anette Maria Borgund Hansen, RN, Cand Scient San stud, Rigshospitalet, Denmark
Other Study IDs: dura010321
Record Dates: First submitted 2021-03-09; First posted 2021-03-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Dural Tear; Bedrest; Lumbar Spine Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of this study is to assess whether lumbar spine surgery patients with dura rupture differ in symptom prevalence and severity from other lumbar spine surgery patients in the early postoperative phase. This is in order to develop a symptom-specific mobilization algorithm (DURAMOB) that can be used to assess whether patients with dura rupture safe can be mobilized earlier after lumbar back surgery to prevent bed rest complications

DETAILED DESCRIPTION:
Accidental dura rupture is a complication of lumbar spine surgery, with an incidence of 2-18% which can cause cerebrospinal fluid leakage leading to symptoms such as postural headache, photosensitivity, tinnitus, infection, and pseudomeningocele. Traditionally, the condition is treated with postoperatively flat bed rest ranging from 0-72 hours, entailing an increased risk of complications due to bed rest. There is inconsistency in the length of prescribed flat bed rest for these patients, and no consensus exists nationally or internationally. The prescription of flat bed rest is generally made by the surgeons based on their clinical experience.

This quality development project in the clinimetric field aims to develop an assessment tool (Duramob) of perioperative symptoms prevalence and severity in lumbar spine surgery patients with and without dura rupture in the early postoperative phase.

Data is based on clinical auditing comprising a consecutive samples of patients in collaboration with " Center for Rheumatology and Spine Diseases", Rigshospitalet-Glostrup, Denmark.

The Duramob instrument will be developed as an evidence-based algorithm for assessing the potential need for postoperatively restrictive bedrest after dura rupture, - and subsequently to be implemented in clinical perioperative practice. Further scientific testing will following be carried out in a feasibility study and / or as a Randomized Controlled Trial.

This initial study will generate observational evidence investigating the first steps towards establishing a safe mobilisation regime for patients with surgical dura rupture. Ultimately, we seek to avoid unnecessary bedrest and complications derived from perioperative immobilization. Data will be protected in a local clinical database RedCap hosted by the Capital Region Data Management system and follows GDPR regulations. The department leadership approved the project and the local ethical Committee' waived the need for approval.

ELIGIBILITY:
Inclusion Criteria:

Lumbar surgery patients age >18 years

-

Exclusion Criteria:

Trauma surgery Cancer surgery lumbar fusion surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lumbar surgery with and without peroperative accidential dural lesion
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Dura rupture symptom severity | 9 month
  To asses whether symptoms or compound of symptoms differ in patients with or without dura rupture in stand up up position 6 and 24 hours after lumbar surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Glostrup, Glostrup Municipality, Denmark